CLINICAL TRIAL: NCT07194772
Title: The Effects of NAtural Sugars, REfined Sugars, and LOw-Calorie Sweeteners on Postprandial Glycemic Responses and Mechanistic Pathways Under Real-World Conditions
Brief Title: Sucralose and Glucose Metabolism in Young Healthy Adults
Acronym: NARELO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-04-20-5636; GR005077 (Other Grant/Funding Number: Faculty of Health Sciences, University of Ottawa)
Record Dates: First submitted 2025-09-18; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Glucose Intolerance; Glucose and Insulin Response; Glucose Homeostasis; Low-grade Inflammation; Intestinal Permeability; Gut Microbiota Diversity and Composition; Gut Microbiota Modulation; Gut Microbiota Dysbiosis; Gut Microbiota; Gut Microbiota Dysbiosis and Nutrition; Insulin Resistance; Insulin Sensitivity/Resistance; Insulin Sensitivity
Keywords: low-calorie sweeteners; sucralose; natural sugars; fruit juice; refined sugars; sugar-sweetened beverages; LCS; SSB; non-nutritive sweeteners; sugar substitutes; gut microbiota; low-calorie sweeteners and gut microbiota; low-calorie sweeteners and glycemic responses; sucralose and gut microbiota; sucralose and glycemic responses
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance | interventions — SSB protein, human

STUDY DESIGN:
Intervention Model Description: randomized parallel-group design stratified by sex
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sucralose-sweetened beverages (low-calorie sweetener) (Experimental)
  Interventions: Other: Low-calorie sweeteners (LCS)
- Sugar-sweetened beverages (refined sugars) (Experimental)
  Interventions: Other: Refined sugars (SSB)
- Natural fruit juice (natural sugars) (Experimental): 100% natural orange juice
  Interventions: Other: Natural sugars (FJ)

INTERVENTIONS:
Other: Low-calorie sweeteners (LCS) — Consumption of sucralose-sweetened beverages (LCS) using doses and formulations reflecting real-world conditions.
  Individualized dose equivalent volume (mL) to SSB group. Average dose received of 150 mg (±30 mg) of pure sucralose per day (2.00 ± 0.23 mg/Kg BW) among participants, which is below Acceptable Daily Intake for sucralose (5 mg/Kg BW/day). LCS matched for sweetness to SSB based on the manufacturer's information.
  Arms: Sucralose-sweetened beverages (low-calorie sweetener)
Other: Refined sugars (SSB) — Consumption of sugar-sweetened beverages (SSB) using doses and formulations reflecting real-world conditions.
  Individualized dose of 15% Ereq representing estimated free sugars consumption in Canada. SSB matched total free sugar concentration of 100% natural orange juice (FJ).
  Arms: Sugar-sweetened beverages (refined sugars)
Other: Natural sugars (FJ) — Consumption of natural fruit juice (100% natural orange juice) using doses and formulations reflecting real-world conditions.
  Individualized dose of 15% Ereq representing estimated free sugars consumption in Canada.
  Arms: Natural fruit juice (natural sugars)

SUMMARY:
This study aimed to investigate the effects of a three-week consumption of sucralose-sweetened beverages (low-calorie sweetener) on postprandial glycemic responses in healthy adults, compared with sugar-sweetened beverages under real-world conditions. In brief, postprandial glycemic responses are used as an indicator of how your body manages blood sugar levels after consuming glucose. To explore potential mechanisms underlying any observed changes in postprandial glycemic responses, we further investigated potential alterations in gut microbiota composition and functionality, as well as plasmatic biomarkers of intestinal permeability and systemic low-grade inflammation. Finally, this project explored whether free sugars derived from a natural source (100% natural fruit juice) elicit metabolic responses that differ from those of refined sugars.

Participants visited the laboratory for a preliminary screening session to assess eligibility prior to being randomly assigned to one of the three experimental groups consuming either sucralose-sweetened beverages (LCS), sucrose-sweetened beverages (SSB), or 100% natural fruit juice (FJ) at dosage approximating real-world consumption over three weeks. Participants underwent two experimental sessions (duration of 3 hours each) at the beginning and completion of the study as outlined below.

DETAILED DESCRIPTION:
PRELIMINARY SESSION (duration of 2h15) :

To determine eligibility, participants were asked to undergo a fasted in-person preliminary session during which the following measures were taken: height, weight, waist circumference, blood pressure, fasting blood glucose (using a glucometer with a capillary blood droplet collected on the fingertip) and answers to two food questionnaires related to dietary habits and food cravings. Upon confirmation of eligibility, participants were offered to continue the preliminary session and informed consent was obtained. Resting metabolic rate (used to determine daily energy needs) was measured using indirect calorimetry. To do so, participants wore a mask that covered their nose and mouth while lying down, awake and motionless for 30 minutes. Lastly, participants received essential information to prepare for their participation in the study. These included specific dietary instructions to follow during the 7-day pre-intervention period and for the duration of the study protocol as well as instructions on proper collection methods of stool samples at home. Specifically, a small quantity of stool samples (2 tubes of 10 mL each) was collected at the beginning and at the end of the study. Participants were asked to transport their frozen stool samples to our research facility at both of their experimental sessions using provided collection materials.

FIRST EXPERIMENTAL SESSION (duration of 3h00) :

The baseline experimental session was scheduled after a 7-day pre-intervention period, marking the beginning of the three-week study. Participants were asked to arrive at the laboratory around 7h30 AM following a 12-hour overnight fast, which began after consuming a standardized meal provided the evening before. Participants were asked to bring their first frozen stool sample (collected at home) to the laboratory as outlined above.

The following tests and procedures were performed :

* Body measurements: height, weight, and waist circumference were measured.
* Blood pressure: blood pressure was measured using an automatic sphygmomanometer, the same kind of equipment used by family physician.
* Body composition: body composition (bone density, lean and fat body mass) was measured using dual energy X-ray absorptiometry (DXA). Participants lied down on an examination table, fully clothed, while a low intensity X-ray scanned the entire body for the duration of five to ten minutes. The radiation level for each DXA scan is lower than the exposition during a transcontinental airplane flight.
* Oral glucose tolerance test (blood samples): An intravenous catheter was placed into the anti-cubital vein in the participants' forearm by certified personnel. This involves the insertion of a needle into a vein through which a small, flexible plastic tubing (catheter) is placed. The needle is then removed, leaving the tubing taped in place. This method allowed us to take blood draws throughout without the need for multiple venous punctures. A fasting 12mL blood sample was drawn immediately after insertion. Then, participants were given 5 minutes to drink a solution containing 75g of glucose. Blood draws of 12 mL each were collected at 30, 60, 90 and 120 min following the ingestion of the glucose solution. Plasma concentrations of glucose and insulin were measured to evaluate glucose homeostasis and insulin sensitivity. Plasmatic biomarkers of intestinal permeability and systemic low-grade inflammation were measured in fasting samples. A total of ~60mL of blood was collected for this procedure, which is a minimal amount. In comparison, a regular blood donation is around 470mL of blood. Participants drank water ad libitum throughout the session. A light snack was provided before the participant was sent home.

Study beverages :

Participants left the first experimental session with a one-week supply of study beverages corresponding to their randomly assigned group : sucralose-sweetened beverages (LCS), sucrose-sweetened beverages (SSB), or 100% natural fruit juice (FJ). Study beverages were designed to realistically reflect commercially available options, and the daily dose was personalized based on each participant's energy needs to simulate real-world intake. Study beverages were provided frozen in a cooler bag, and participants were instructed to consume one bottle per day (divided into three doses with meals) and to keep the bottles refrigerated. On weeks 2 and 3, participants returned to the laboratory to pick up their weekly supply and drop off used bottles (two visits total).

SECOND EXPERIMENTAL SESSION (duration of 3h00) :

A second experimental session was scheduled on day 22, that is after consuming study beverages for three weeks. The post-experimental sessions marked the end of the study. The same tests and procedures that occurred during the first experimental session were repeated.

TIMELINE SUMMARY :

* Preliminary session
* 7-day pre-intervention period
* Two small stool samples collected at home
* Day 0 : First experimental session including blood draws
* 21 days of consuming study beverages (two visits for pick-up and return of weekly supplies)
* Two small stool samples collected at home
* Day 22 : Second experimental session including blood draws

ELIGIBILITY:
INCLUSION CRITERIA included ages 18-35 y, body mass index (BMI) between 18.0 and 34.9 kg/m2, waist circumference < 102cm (men) and < 88cm (women) and a self-reported stable weight during the prior 6 months (+ or - 2kg) of beginning the study.

Additional Considerations related to the menstrual cycle and the use of hormonal contraceptives : All women who participated in this study were premenopausal. Recognizing the crucial importance of including women in our study while ensuring the highest quality data, additional considerations were applied to meet inclusion criteria: Women using no form of hormonal contraception or using copper intrauterine device (IUD) required to report having a regular menstrual cycle to be included; Women using anovulants (birth control pills) were advised to take their daily anovulant continuously for a period of 28 days to ensure stable hormone levels throughout the study (informed consent was obtained). Oral contraceptives release a low and stable daily amount of progestins, which were reported to have minor or no effects on glycemic responses of pre-menopausal women in a recent meta-analysis38; Women using hormonal contraception such as hormonal IUD and subdermal contraceptive implant were included regardless of their menstrual cycle. Like anovulants, hormonal IUD release a low and stable amount of a progestin (levonorgestrel) into the uterus, therefore preventing periodic fluctuations in hormonal levels during the menstrual cycle. Since Levonorgestrel was included as one of the progestins in the aforementioned meta-analysis38, it was therefore assumed that HIUD would also not have a significant impact on glycemic responses, especially as its effect is local rather than systemic; Women using medroxyprogesterone acetate injections (Depo-Provera shot) were excluded given the pro-inflammatory effects associated with high doses of progestin; Women experiencing pregnancy or lactation were excluded.

EXCLUSION CRITERIA consisted of prediabetes (fasting glucose ≥ 6.1 mmol/L), diabetes (fasting glucose ≥ 7.0 mmol/L), hypertension (> 140/90 mmHg), personal medical history for dyslipidemias (including hypercholesterolemia and hypertriglyceridemia), and surgery for weight loss. In addition, individuals who smoke tobacco (including vaping), habitually ingest >2 alcoholic beverages/day, use cannabis or cannabis-derived products >1 time/month , exercise >3.5 h/week at a level more vigorous than walking, or use thyroid, lipid-lowering, glucose-lowering, antihypertensive, antidepressant/antianxiety, antibiotics in the prior 3 months or weight-loss medications were excluded. Finally, individuals susceptible to exhibit clinically relevant levels of food cravings as indicated by a score > 50 on the Food Cravings Questionnaire - Trait reduced (FCQ-T-r)36, were also excluded. FCQ-T-r (15 items) is a validated questionnaire37 that assesses four factors: (1) preoccupation with food (i.e., obsessive thought about food and eating), (2) loss of control (i.e., difficulty regulating eating behavior when exposed to food cues), (3) positive outcome expectancy (i.e., believing eating to be positively reinforcing), and (4) emotional craving (i.e., tending to crave food when experiencing negative emotion).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Postprandial Glycemic Responses | 3 weeks
  Postprandial Glycemic Responses (plasma glucose concentrations) were assessed using a 2-hour 75g Oral Glucose Tolerance Test (OGTT) at baseline (day 0) and post-intervention (day 22)

SECONDARY OUTCOMES:
Change from Baseline in Postprandial Insulinemic Responses | 3 weeks
  Postprandial Insulinemic Responses (plasma insulin concentrations) were assessed using a 2-hour 75g Oral Glucose Tolerance Test (OGTT) at baseline (day 0) and post-intervention (day 22)
Change from Baseline in Plasmatic Biomarkers of Intestinal Permeability | 3 weeks
  Plasmatic Biomarkers of Intestinal Permeability (Zonulin, LBP) were assessed in fasting plasma samples at baseline (day 0) and post-intervention (day 22)
Change from Baseline in Plasmatic Biomarkers of Systemic Low-grade Inflammation | 3 weeks
  Plasmatic biomarkers of systemic low-grade inflammation (IL-6, TNF-a, CRP) were assessed in fasting plasma samples at baseline (day 0) and post-intervention (day 22)
Change from Baseline in Fecal Concentrations of Short-Chain Fatty Acids and Branched-Chain Fatty Acids | 3 weeks
  Fecal Concentrations of Short-Chain Fatty Acids and Branched-Chain Fatty Acids were measured at baseline (day 0) and post-intervention (day 22). Two serial stool samples were collected on separate days within the three days preceding both the baseline and post-experimental sessions.
Change from Baseline in Alpha-diversity and Beta-diversity of the Fecal Microbiota | 3 weeks
  Alpha-diversity and Beta-diversity of the Fecal Microbiota were measured at baseline (day 0) and post-intervention (day 22). Two serial stool samples were collected on separate days within the three days preceding both the baseline and post-experimental sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Behavioural and Metabolic Research Unit, School of Human Kinetics, Faculty of Health Sciences, University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All de-identified individual participant data that underlie the results reported in the publication, including participants characteristics, outcomes measures (i.e., glycemic-insulinemic responses, plasmatic biomarkers of intestinal permeability and low-grade inflammation as well as microbiota outcomes) and relevant covariates will be shared. Supporting documents such as the study protocol and statistical analysis plan will also be available upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 1 year after publication and available for 2 years.
Access Criteria: Available to qualified researchers upon request (via institutional repository or upon request to the PI) and approval of a research proposal and data sharing agreement.